CLINICAL TRIAL: NCT00223340
Title: Diabetes and Cardiovascular Risks in Primary Care
Brief Title: The ABC Planning Study: Diabetes and Cardiovascular Risks in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single
Other Study IDs: 1 R34 DK 067300-1A1 [NIDDK]; 1 R34 DK 067300-1A1 [NIDDK]; 1R34DK067300 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Diabetes
Keywords: patient activation; primary care; diabetes; cardiovascular risk
MeSH Terms: conditions — Diabetes Mellitus; Patient Participation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Patient Activation and Diabetes Registry

SUMMARY:
The purpose of this pilot study is to collect preliminary information about the best way to implement an intervention to reduce the risks of heart disease and stroke.

DETAILED DESCRIPTION:
This study has two types of interventions. The clinics and patients are randomly assigned to either a control or intervention group. All clinics have both control and intervention patients. In the clinic intervention, we help doctors monitor patient information about the risk factors of heart disease and stroke. In the patient intervention, we contact patients by phone to discuss these risk factors before their doctor visits.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be diagnosed with diabetes for at least 12 months.
* Patient must be with current physician for at least 12 months.
* Study staff must be able to reach patient by telephone.

Exclusion Criteria:

* Pregnant women are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2005-03; Primary Completion 2007-06 (Actual); Study Completion 2007-06

PRIMARY OUTCOMES:
Document changes made to study procedures to better implement this study's interventions that are designed to reduce risks of heart disease and stroke

SECONDARY OUTCOMES:
Patient Outcome Measures: Hemoglobin A1c (HbA1c), lipids (low-density lipoprotein [LDL] non-high-density lipoprotein [HDL] triglycerides), blood pressure
Patient assessed health status, diabetes self-care activities and knowledge of cardiovascular (CV) risk factors
Physician Outcome Measures: Physician knowledge, attitude and readiness to change practice; Physician-level measure of patient-centeredness of encounter and interpersonal communication
Assessment of Chronic Illness Care (ACIC) Surveys

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Parchman, MD, MPH, Principal Investigator — Univ. of Texas Health Science Center at San Antonio
Locations (1):
- The University of Texas Health Science Center at San Antonio (Texas), San Antonio, Texas, United States